CLINICAL TRIAL: NCT07185724
Title: Balancing Comfort and Success: Post-retrieval Ketorolac in Fresh Embryo Transfers
Brief Title: Ketorolac Use and Fresh Embryo Transfer Outcomes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jessica D. Kresowik (Other)
Responsible Party: Sponsor-Investigator, Jessica D. Kresowik, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202505454
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Infertility (IVF Patients); Infertility Treatment; Post-op Pain; Fresh Embryo Transfer; Oocyte Retrieval and Post Operative Pain Control
Keywords: IVF; post operative pain control; oocyte retrieval; fresh embryo transfer; ketorolac; toradol; implantation rate; live birth rate; miscarriage rate
MeSH Terms: conditions — Infertility; Pain, Postoperative | interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, investigator, IVF provider, nursing team, and all members involved in assessing outcomes will be blinded. Patient will be under anesthetic influence and be unaware of medication administration. Recovery nurse and surgeon will not be aware or informed of treatment arm.
  Anesthesia will be unblinded but will not inform any other members of the medical team whether or not patient received ketorolac.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV Ketorolac (Experimental): Participants randomized to this arm will receive 30mg IV Ketorolac at the conclusion of their oocyte retrieval.
  Interventions: Drug: Ketorolac 30 mg IV
- No IV Ketorolac (No Intervention): Participants randomized to this arm will not receive IV Ketorolac at the conclusion of their oocyte retrieval.

INTERVENTIONS:
Drug: Ketorolac 30 mg IV — We will be evaluating the effect of post-oocyte retrieval ketorolac administration on clinical outcomes in fresh embryo transfer cycles.
  Arms: IV Ketorolac

SUMMARY:
Ketorolac is a medication often used to relieve pain after surgery. In the past, infertility doctors have been cautious about using ketorolac after egg retrieval for patients planning a fresh embryo transfer (usually done 5 days later). The concern was that ketorolac might increase the risk of bleeding or reduce the chances of the embryo implanting in the uterus. This concern comes from how ketorolac works-it blocks certain chemicals in the body (like prostaglandins and thromboxane) that help with blood clotting and play a role in early pregnancy.

However, a large review of past studies found no real evidence that ketorolac increases bleeding risk. In fact, ketorolac is now routinely used for pain relief in IVF cycles where embryos are frozen and not transferred right away. More recent studies from Boston and Chapel Hill have shown that ketorolac provides better pain control and does not appear to harm IVF outcomes, even when embryos are transferred fresh (within the same cycle).

Despite these encouraging findings, many IVF clinics still avoid using ketorolac during fresh cycles because of the theoretical concerns. That's why we need stronger, higher-quality research.

This study aims to fill that gap by conducting a double-blind randomized controlled trial to find out whether giving ketorolac through an IV after egg retrieval affects important IVF outcomes-especially the chance of implantation and live birth-in patients undergoing fresh embryo transfers. Patients who choose to join the study will randomly be placed into one of two groups. One group will get ketorolac (a pain medicine) after an IVF egg retrieval. The other group will not get ketorolac after egg retrieval. Everything else in their IVF care will stay the same as it normally would.

Primary outcome will be implantation rate following fresh embryo transfers in patients receiving ketorolac (30mg IV) vs no ketorolac for post-retrieval analgesia.

Secondary outcomes will include pain scale, narcotics required, time to discharge, need for evaluation w/in 24 hours for pain/bleeding, clinical pregnancy rates, miscarriage rates, and live birth rates following fresh embryo transfers in patients receiving ketorolac vs no ketorolac for post-retrieval analgesia.

DETAILED DESCRIPTION:
Study Design: double-blind randomized controlled trial Intervention: Ketorolac (30mg intravenous) administration in the immediate post-operative period prior to leaving the procedure room and while patient is still under sedation

Allocation method: 1:1 statistician generated block randomization (blocks of 2, 4, and 6). Patients will be randomized immediately following consent and enrollment.

Materials and Methods: Patients undergoing an IVF autologous cycle at our institution where the female patient is planning on proceeding with a fresh embryo transfer 5 days following ultrasound guided oocyte retrieval will be recruited. Patients may undergo any of our standard controlled ovarian hyperstimulation protocols.

On the day of egg retrieval patients will:

* Sign the consent and be randomly assigned to one of two groups (usual care plus ketorolac OR usual care without ketorolac).
* At the end of the retrieval procedure while the patient is still under sedation, the anesthesiology team will administer either usual care plus ketorolac OR usual care without ketorolac through the pre-existing IV line.

Patients IVF care will otherwise remain the same as planned, including:

* Monitoring in the recovery area as per standard protocol
* Embryo transfer on day 5 post-retrieval

Investigators will continue to review and collect data from patients' medical records for up to 45 weeks. This will include demographic and medical information, including, but not limited to:

* age, medical diagnosis, physical exam findings such as height and weight, laboratory testing, and ultrasound results
* reproductive history including how long patients have been trying to conceive, infertility diagnoses, outcomes of past pregnancies, outcomes of prior infertility evaluation and treatments
* the types and doses of medications used, types of infertility treatments used, and information about patients' treatment cycles. Treatment cycle information will include, but is not limited to:
* response to ovarian stimulation,
* sperm count,
* embryo development and quality,
* any post-retrieval evaluations for pain and/or bleeding, and
* whether or not a pregnancy resulted.
* narcotic use during recovery, and time to discharge
* Outcomes from the fresh embryo transfer following retrieval. If patients conceive a pregnancy, then investigators will follow the pregnancy through its resolution. Investigators will collect information about patients:
* pregnancy hormone levels,
* confirmation or pregnancy ultrasound findings,
* information on implantation, clinical pregnancy, miscarriage, and live births.

ELIGIBILITY:
Inclusion Criteria:

* IVF utilizing autologous oocytes and all sperm sources
* IVF cycles utilizing ICSI and standard insemination
* Plan to transfer embryo on day 5
* BMI below 50

Exclusion Criteria:

-allergies or medical contraindications to NSAIDs

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-08 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Implantation Rate | From enrollment to the time of confirmation of pregnancy ultrasound at ~6 weeks post-oocyte retrieval (with or without administration of IV Ketorolac) .
  Implantation rate following fresh embryo transfers in patients receiving ketorolac vs no ketorolac for post-retrieval analgesia. We define implantation rate as the proportion of transferred embryos which resulted in fetal heartbeat seen on ultrasound per patient.

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | From enrollment to the time of confirmation of pregnancy ultrasound at ~6 weeks post-oocyte retrieval (with or without administration of IV Ketorolac) .
  Clinical pregnancy rate is defined as the proportion of patients who had an embryo transfer which resulted in a pregnancy confirmed by an increasing level of human Chorionic Gonadotropin (hCG) and the presence of a gestational sac detected by ultrasound.
Miscarriage Rate | From date of enrollment through first documented instance of miscarriage up to 40 weeks.
  Miscarriage rate is defined as the percentage of patients with miscarriage after a clinical pregnancy.
Live Birth Rate | From enrollment to the end of pregnancy (~40 weeks) resulting from fresh embryo transfer following the oocyte retrieval in which patient received IV Ketorolac or no IV Ketorolac.
  Live birth rate is defined as percentage of patients who had a transfer which resulted in a live birth.
Post-operative Pain | From enrollment until the time of discharge from oocyte retrieval (~2.5 hours).
  In the immediate post-operative period, pain will be assessed per standard practice using the visual analog scale. The visual analog scale is used to assess pain on a scale of 0 to 10 with 0 being no pain and 10 being worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- UI Health Care Center for Advanced Reproductive Care, Iowa City, Iowa, United States

REFERENCES:
- [Background] Mesen TB, Kacemi-Bourhim L, Marshburn PB, Usadi RS, Matthews M, Norton HJ, Hurst BS. The effect of ketorolac on pregnancy rates when used immediately after oocyte retrieval. Fertil Steril. 2013 Sep;100(3):725-8. doi: 10.1016/j.fertnstert.2013.04.048. Epub 2013 May 28. PMID 23721715
- [Background] Gobble RM, Hoang HLT, Kachniarz B, Orgill DP. Ketorolac does not increase perioperative bleeding: a meta-analysis of randomized controlled trials. Plast Reconstr Surg. 2014 Mar;133(3):741-755. doi: 10.1097/01.prs.0000438459.60474.b5. PMID 24572864
- [Background] Waljee JF, Li L, Brummett CM, Englesbe MJ. Iatrogenic Opioid Dependence in the United States: Are Surgeons the Gatekeepers? Ann Surg. 2017 Apr;265(4):728-730. doi: 10.1097/SLA.0000000000001904. No abstract available. PMID 27429023

DOCUMENTS (1):
  • Informed Consent Form (2025-08-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT07185724/ICF_000.pdf